CLINICAL TRIAL: NCT00450034
Title: Impact of Optimization of Drug Treatment of Elderly Admitted in 4 Acute Geriatric Wards : Randomized Trial
Brief Title: Optimization of Drug Treatment in Hospitalized Elderly (OMAGE)
Acronym: OMAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P060247
Record Dates: First submitted 2007-03-19; First posted 2007-03-21 (Estimated); Last update posted 2011-12-01 (Estimated); Status verified 2007-03

CONDITIONS: Global Medical Assessment of Elderly Frail Patients
Keywords: Frail Elderly; Patient Education; Drug optimization; Underuse; Vulnerable; Drug related hospitalization; Medical intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Procedure: drug - oriented multifaceted intervention

INTERVENTIONS:
Procedure: drug - oriented multifaceted intervention — oriented multifaceted intervention

SUMMARY:
A randomized trial has been designed to determine if this complex intervention can significantly decrease the risk of unplanned readmissions in this very elderly population, compared with usual care.

DETAILED DESCRIPTION:
Drug treatment in elderly is not yet optimal. 20 to 30% of admissions of elderly aged over 80 are related to drug problems, most of them being preventable. To decrease drug related hospitalizations need iatrogenic prevention, compliance improvement, and underuse decrease. A multifaceted intervention has been designed, included three dimensions : 1/ drug optimization 2/ patient and/or caregiver education and 3/ better coordination with home health professionals before discharge.

A randomized trial has been designed to determine if this complex intervention can significantly decrease the risk of unplanned readmissions in this very elderly population, compared with usual care.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized as a matter of urgency in unity(unit) of geriatrics acute
* Patients of more than 70 years old
* Hospitalization in the Unity(Unit) of Geriatrics foreseen(planned) superior acute in 5 days
* enlightened assent writing and signed
* preliminary medical examination

Exclusion Criteria:

* Patients in scheduled(programmed) hospitalization
* Patient in palliative care
* Patient whose vital forecast is engaged(opened) in 3 months
* Patient already include during a previous hospitalization Patient already included in a study concerning the therapeutic care
* Followed medical impossible (refusal of care, absence of alive regular, patient doctor abroad)
* not membership to a regime of Social Security or CMU
* Patient not speaking French

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 665 (Actual)
Dates: Start 2007-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Rate of unplanned readmissions, including emergency consultations, | during the study

SECONDARY OUTCOMES:
Mortality at 6 months, | at 6 months
delay before readmission, | before readmission
number of drug events related readmissions. | readmissions
Data collected at 3 and 6 months | at 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie LEGRAIN, MD,PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Chu Bichat Claude Bernard, Paris, France

REFERENCES:
- [Result] Legrain S, Tubach F, Bonnet-Zamponi D, Lemaire A, Aquino JP, Paillaud E, Taillandier-Heriche E, Thomas C, Verny M, Pasquet B, Moutet AL, Lieberherr D, Lacaille S. A new multimodal geriatric discharge-planning intervention to prevent emergency visits and rehospitalizations of older adults: the optimization of medication in AGEd multicenter randomized controlled trial. J Am Geriatr Soc. 2011 Nov;59(11):2017-28. doi: 10.1111/j.1532-5415.2011.03628.x. Epub 2011 Sep 27. PMID 22091692